CLINICAL TRIAL: NCT04353284
Title: The Effect of Camostat Mesylate on COVID-19 Infection in Ambulatory Patients: An Investigator-Initiated Randomized, Placebo-Controlled, Phase IIa Trial
Brief Title: Camostat Mesylate in COVID-19 Outpatients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000027971
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Camostat mesylate (Experimental): Camostat mesylate 200mg taken 7 days.
  Interventions: Drug: Camostat Mesilate
- Placebo (Placebo Comparator): Placebo taken for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Camostat Mesilate — Camostat mesilate 200mg taken orally, 4 times daily, for 7 days.
  Other Names: Fiopan, Camostat Mesylate
  Arms: Camostat mesylate
Other: Placebo — Placebo taken orally, 4 times daily, for 7 days.
  Arms: Placebo

SUMMARY:
The rationale of the present clinical trial is that an orally available drug given to outpatients that could reduce the viral burden in the upper respiratory tract could forestall complications of SARS-CoV-2 infection and reduce transmission from one infected individual to another.

DETAILED DESCRIPTION:
The study is designed as a double-blind randomized controlled clinical trial to test the hypothesis that camostat mesylate, a serine protease inhibitor shown to inhibit SARS-COV-2 replication in vitro, inhibits SARS-COV-2 replication in early stage, laboratory-confirmed, COVID-19 ambulatory patients.

Camostat mesylate, a serine protease inhibitor used primarily for treating postoperative reflux esophagitis and for acute exacerbations of chronic pancreatitis. This drug, with more than 15 years clinical experience in Japan with a very safe clinical track record, will be studied as a repurposed drug based on published in vitro virus inhibition data and in vivo protective effects in a mouse model of SARS.

The primary objective of this study is to determine whether camostat mesylate reduces SARS-COV-2 viral load in early COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled within 3 days of being notified of their first positive COVID-19 test result.
* Evidence of a recent active COVID-19 infection, as evidenced by the positive test results being associated with at least one COVID-19-compatible symptom such as fever, upper respiratory symptoms, cough, chills, loss of taste/smell, etc.(see COVID-19-PRO symptom score sheet), or a recent high-risk exposure to COVID-19
* Provision of informed consent.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Diagnosed with COVID-19 within past 3 days and not exhibiting manifestations requiring hospitalization such as extreme shortness of breath or severe prostration. Nurses at the study site will assess such severe conditions requiring hospitalization, which would preclude enrollment.
* Ability to take oral medication and be willing to adhere to the camostat mesylate regimen.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of the camostat mesylate administration.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration.
* English and Spanish speaking subjects as well as patients speaking any language for which we can find appropriate translators will be enrolled. A short form with interpretation will be used for anyone speaking a language for which a translated informed consent form is not currently available in accordance with local site IRB policies, including developing certified translations as necessary.

Exclusion Criteria:

* Presence of COVID-19 disease manifestations that would require referral for consideration of hospitalization.
* A previous positive COVID-19 test reported more than 7 days before, which would indicate likelihood of non-culturable, nonreplicating virus.
* A positive COVID-19 test without a known recent exposure that would indicate an active infection, hence an unknown chance of non-culturable, non-replicating virus being present (i.e., asymptomatic COVID-19 infection of unknown duration).
* Pregnancy or lactation.
* Known allergic reactions to components of camostat mesylate.
* With regard to inclusion or exclusion of women of child-bearing potential, women who report that they know they are pregnant are excluded. All women of child-bearing potential who test positive for pregnancy by urine test at first visit are excluded. A day 14 followup blood pregnancy test will be done on appropriate enrolled women (i.e. those who had a negative urine pregnancy test on day 0 for further safety assessment ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Chupp, M.D., Principal Investigator — Director, Yale Center for Asthma and Airways Disease (YCAAD); Joseph Vinetz, M.D., Principal Investigator — Professor, Section of Infectious Diseases: Department of Internal Medicine
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kosinsky Y, Peskov K, Stanski DR, Wetmore D, Vinetz J. Semi-Mechanistic Pharmacokinetic-Pharmacodynamic Model of Camostat Mesylate-Predicted Efficacy against SARS-CoV-2 in COVID-19. Microbiol Spectr. 2022 Apr 27;10(2):e0216721. doi: 10.1128/spectrum.02167-21. Epub 2022 Apr 12. PMID 35412356
- [Derived] Chupp G, Spichler-Moffarah A, Sogaard OS, Esserman D, Dziura J, Danzig L, Chaurasia R, Patra KP, Salovey A, Nunez A, May J, Astorino L, Patel A, Halene S, Wang J, Hui P, Patel P, Lu J, Li F, Gan G, Parziale S, Katsovich L, Desir GV, Vinetz JM. A Phase 2 Randomized, Double-Blind, Placebo-controlled Trial of Oral Camostat Mesylate for Early Treatment of COVID-19 Outpatients Showed Shorter Illness Course and Attenuation of Loss of Smell and Taste. medRxiv [Preprint]. 2022 Jan 31:2022.01.28.22270035. doi: 10.1101/2022.01.28.22270035. PMID 35132421

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Camostat Mesylate | Placebo
Started | 35 | 35
Completed | 33 | 34
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat Mesylate | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (14.6) | 44.1 (12.0) | 44.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 28 | 29 | 57
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in SARS-COV-2 Viral Load
Description: To determine whether camostat mesylate reduces SARS-COV-2 viral load (N Gene) in early COVID-19 disease, change from day 0 to day 4 in respiratory (oropharyngeal swab RT-PCR) log10 viral load will be assessed.
Time Frame: 5 days (day 0 to day 4)
Population: Intention to treat, baseline is pooled across treatment arms in the mixed models analysis as Day 0/Baseline data were collected prior to treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
log10 copies/mL
  Day 0 | 6.5 [6.0 to 6.9] | 6.5 [6.0 to 6.9]
  Day 4 | 4.4 [3.8 to 5.1] | 3.7 [3.0 to 4.3]
  Change (Day 4 - Day 0) | -2.0 [-2.6 to -1.5] | -2.8 [-3.3 to -2.2]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; This analysis compares the change from baseline between treatment arms; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = 0.74, 95% CI 2-sided [-0.03 to 1.51]

2. Secondary Outcome: Change in SARS-COV-2 Viral Load
Description: To determine whether camostat mesylate reduces SARS-COV-2 viral load (N Gene) in early COVID-19 disease, change from day 0 to day 2 in respiratory (oropharyngeal swab RT-PCR) log10 viral load will be assessed.
Time Frame: 3 days (day 0 to day 2)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
log10 copies/mL | -1.2 [-1.8 to -0.6] | -1.3 [-1.8 to -0.7]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.87, Mixed Models Analysis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.70 to 0.83]

3. Secondary Outcome: Change in SARS-COV-2 Viral Load
Description: To determine whether camostat mesylate reduces SARS-COV-2 viral load (N Gene) in early COVID-19 disease, change from day 0 to day 6 in respiratory (oropharyngeal swab RT-PCR) log10 viral load will be assessed.
Time Frame: 7 days (day 0 to day 6)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
log10 copies/mL | -3.6 [-4.5 to -2.8] | -3.9 [-4.7 to -3.0]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.94 to 1.4]

4. Secondary Outcome: Number of Participants With Change in Positive COVID-19 Status
Description: Change in risk for a positive COVID-19 test at day 6 after enrollment (day 0) will be assessed by analyzing the proportion of positive cases in each study arm.
Time Frame: 7 days
Population: Intention to treat analysis using all participants with data at 7 days, 14 days and 28 days. The model excluded those with baseline data only (1 Camostat, 1 Placebo). Participants with valid data are presented at 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 34 | 34
Participants
  Nasopharyngeal Swab Samples: number analyzed (Participants) | 22 | 25
  Nasopharyngeal Swab Samples: Positive | 17 | 18
  Nasopharyngeal Swab Samples: Negative | 5 | 7
  Saliva RT-PCR: number analyzed (Participants) | 22 | 25
  Saliva RT-PCR: Positive | 14 | 21
  Saliva RT-PCR: Negative | 8 | 4
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Nasopharyngeal Swab Samples analyzed; Test type: Superiority; p = 0.71, GEE; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.33 to 5.09]
Statistical Analysis 2: Comparison: Camostat Mesylate vs Placebo; Saliva RT-PCR samples analyzed; Test type: Superiority; p = 0.17, GEE; Within subject correlation is controlled by specifying a compound symmetry R-side structure in the model; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.11 to 1.47]

5. Secondary Outcome: Number of Participants With Change in Positive COVID-19 Status
Description: Change in risk for a positive COVID-19 test at day 13 after enrollment (day 0) will be assessed by analyzing the proportion of positive cases in each study arm.
Time Frame: 14 days
Population: Intention to treat analysis using all participants with data at 7 days, 14 days and 28 days. The model excluded those with baseline data only (1 Camostat, 1 Placebo). Participants with valid data are presented at 14 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 34 | 34
Participants
  Nasopharyngeal Swab Samples: number analyzed (Participants) | 33 | 33
  Nasopharyngeal Swab Samples: Positive | 21 | 12
  Nasopharyngeal Swab Samples: Negative | 12 | 21
  Saliva RT-PCR: number analyzed (Participants) | 33 | 32
  Saliva RT-PCR: Positive | 16 | 14
  Saliva RT-PCR: Negative | 17 | 18
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.03, GEE; Within subject correlation is controlled by specifying a compound symmetry R-side structure in the model; Odds Ratio (OR) = 3.05, 95% CI 2-sided [1.12 to 8.26]
Statistical Analysis 2: Comparison: Camostat Mesylate vs Placebo; Saliva RT-PCR samples analyzed; Test type: Superiority; p = 0.68, GEE; Within subject correlation is controlled by specifying a compound symmetry R-side structure in the model; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.47 to 3.23]

6. Secondary Outcome: Change in Positive COVID-19 Status
Description: Number of Participants With Change in Positive COVID-19 Status
Time Frame: 28 days
Population: Intention to treat analysis using all participants with data at 7 days, 14 days and 28 days. The model excluded those with baseline data only (1 Camostat, 1 Placebo). Participants with valid data are presented at 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 34 | 34
Participants
  Nasopharyngeal Swab Samples: number analyzed (Participants) | 32 | 34
  Nasopharyngeal Swab Samples: Positive | 5 | 1
  Nasopharyngeal Swab Samples: Negative | 27 | 33
  Saliva RT-PCR: number analyzed (Participants) | 32 | 34
  Saliva RT-PCR: Positive | 5 | 6
  Saliva RT-PCR: Negative | 27 | 28
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.10, GEE; Within subject correlation is controlled by specifying a compound symmetry R-side structure in the model; Odds Ratio (OR) = 6.28, 95% CI 2-sided [0.70 to 56.60]
Statistical Analysis 2: Comparison: Camostat Mesylate vs Placebo; Saliva RT-PCR samples analyzed; Test type: Superiority; p = 0.87, GEE; Within subject correlation is controlled by specifying a compound symmetry R-side structure in the model; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.25 to 3.23]

7. Secondary Outcome: Change in COVID-19 Symptom Severity
Description: Change of COVID-19 symptom severity from day 0 to day 6 will be assessed with the COVID-19 daily self score tool. Adapted from the FLU-PRO instrument, it consists of 39 items that are answered daily. Items 1-33 are Likert scale questions (rated 0-4) where 0 = not at all and 4 = very much. These items are summed to score the severity of symptoms- where a total score of 132 would indicate the greatest severity of symptoms and a score of 0 would indicate no severity of symptoms. Items 34-38 are also Likert scale questions (rated 0-4) that measure the frequency of specific daily symptoms where 0 = 0 times and 4 = 4 times or more. These items are summed to score the frequency of symptoms- where the highest score for the frequency of symptoms (20) indicates the greatest burden of symptom frequency. The last question (39) asks patients for their highest temperature in Fahrenheit.
Time Frame: Day 0 to Day 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 | 31.5 [27.3 to 35.8] | 31.5 [27.3 to 35.8]
  Day 6 | 12.4 [7.3 to 17.5] | 19.1 [14.0 to 24.1]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -6.6, 95% CI 2-sided [-12.1 to -1.2]

8. Secondary Outcome: Change in COVID-19 Symptom Severity
Description: Change of COVID-19 symptom severity from day 0 to day 14 will be assessed with the COVID-19 daily self score tool. Adapted from the FLU-PRO instrument, it consists of 39 items that are answered daily. Items 1-33 are Likert scale questions (rated 0-4) where 0 = not at all and 4 = very much. These items are summed to score the severity of symptoms- where a total score of 132 would indicate the greatest severity of symptoms and a score of 0 would indicate no severity of symptoms. Items 34-38 are also Likert scale questions (rated 0-4) that measure the frequency of specific daily symptoms where 0 = 0 times and 4 = 4 times or more. These items are summed to score the frequency of symptoms- where the highest score for the frequency of symptoms (20) indicates the greatest burden of symptom frequency. The last question (39) asks patients for their highest temperature in Fahrenheit.
Time Frame: Day 0 to Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 | 31.5 [27.3 to 35.8] | 31.5 [27.3 to 35.8]
  Day 13 | 7.8 [2.5 to 13.2] | 9.9 [4.8 to 15.1]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = -2.1, 95% CI 2-sided [-7.9 to 3.7]

9. Secondary Outcome: Change in COVID-19 Symptom Frequency
Description: Change of COVID-19 symptom frequency score from day 0 to day 6 will be assessed with the COVID-19 daily self score tool. Adapted from the FLU-PRO instrument, it consists of 39 items that are answered daily. Items 34-38 measure the frequency of specific daily symptoms and are also Likert scale questions (rated 0-4) that measure the frequency of specific daily symptoms where 0 = 0 times and 4 = 4 times or more. These items are summed to score the frequency of symptoms- where the highest score (20) indicates the greatest burden of symptom frequency, the lowest possible score (0) indicates no frequency of symptoms.
Time Frame: Day 0 to Day 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 | 5.9 [5.0 to 6.8] | 5.9 [5.0 to 6.8]
  Day 6 | 5.0 [3.9 to 6.2] | 4.1 [3.0 to 5.2]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.4 to 2.3]

10. Secondary Outcome: Change in COVID-19 Symptom Frequency
Description: as for outcome 9
Time Frame: Day 0 to Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Day 0 | 5.9 [5.0 to 6.8] | 5.9 [5.0 to 6.8]
  Day 13 | 2.7 [1.5 to 4.0] | 2.1 [0.9 to 3.2]
Statistical Analysis 1: Comparison: Camostat Mesylate vs Placebo; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.7 to 2.1]

11. Secondary Outcome: Change in Body Temperature
Description: Change of COVID-19 symptom score from baseline to day 6 will be assessed with the COVID-19 daily self score tool. Adapted from the FLU-PRO instrument, it consists of 39 items that are answered daily. Items 1-33 are Likert scale questions (rated 0-4) where 0 = not at all and 4 = very much. These items are summed to score the severity of symptoms- where a total score of 132 would indicate the greatest severity of symptoms and a score of 0 would indicate no severity of symptoms. Items 34-38 are also Likert scale questions (rated 0-4) that measure the frequency of specific daily symptoms where 0 = 0 times and 4 = 4 times or more. These items are summed to score the frequency of symptoms- where the highest score for the frequency of symptoms (20) indicates the greatest burden of symptom frequency. The last question (39) asks patients for their highest temperature in Fahrenheit.
Time Frame: 7 days (Day 0 to Day 6)
Population: Data are presented for those with valid temperature data. Body temperature was not evenly collected at all visits as originally intended.
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 22 | 27
degrees Fahrenheit
  Day 0 | 98.5 (0.8) | 98.3 (0.8)
  Day 6: number analyzed (Participants) | 16 | 19
  Day 6 | 98.0 (1.0) | 98.1 (0.7)

12. Secondary Outcome: Change in Body Temperature
Description: Change of COVID-19 symptom score from baseline to 28 days will be assessed with the COVID-19 daily self score tool. Adapted from the FLU-PRO instrument, it consists of 39 items that are answered daily. Items 1-33 are Likert scale questions (rated 0-4) where 0 = not at all and 4 = very much. These items are summed to score the severity of symptoms- where a total score of 132 would indicate the greatest severity of symptoms and a score of 0 would indicate no severity of symptoms. Items 34-38 are also Likert scale questions (rated 0-4) that measure the frequency of specific daily symptoms where 0 = 0 times and 4 = 4 times or more. These items are summed to score the frequency of symptoms- where the highest score for the frequency of symptoms (20) indicates the greatest burden of symptom frequency. The last question (39) asks patients for their highest temperature in Fahrenheit.
Time Frame: 28 days
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Camostat Mesylate | Placebo
Number analyzed (Participants) | 22 | 27
degrees Fahrenheit
  Day 0 | 98.5 (0.8) | 98.3 (0.8)
  Day 27: number analyzed (Participants) | 13 | 15
  Day 27 | 97.8 (0.5) | 97.7 (0.8)

ADVERSE EVENTS:
Time Frame: Up to 28 days
Arm/Group | Camostat Mesylate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/35
Other Adverse Events (participants affected / at risk) | 3/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camostat Mesylate (N=35) | Placebo (N=35)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camostat Mesylate (N=35) | Placebo (N=35)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04353284/Prot_SAP_000.pdf